CLINICAL TRIAL: NCT07137026
Title: Implementation of Trauma-informed HIV Care With Youth in Memphis, TN
Brief Title: Trauma-informed Care for Youth With HIV in Memphis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-08-1234
Record Dates: First submitted 2025-05-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This is an Interrupted Time Series design study that does not have a control group but rather outcomes are observed based on change between and within individuals from their pre-test scores to their post-test scores, quasi experimentally. There are two arms listed only because one arm is for personnel, which is a training-based intervention, and the other arm is for patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personnel and patients of the clinic (Experimental): This is an interrupted time series where we will compare before and after outcomes based on personnel and patients who receive brief interventions for psychological trauma, comparing personnel wellness outcomes, patient HIV appointment adherence and trauma response outcomes.
  Interventions: Behavioral: Personnel intervention and patients

INTERVENTIONS:
Behavioral: Personnel intervention and patients — The personnel intervention has three components. They are listed above. The patient intervention will include a brief assessment and intervention.
  Other Names: Personnel: Presence 5 for Racial Justice (P5RJ); Personnel: Trauma Stewardship (TS); Personnel: Trauma Resilience (TR); Patient intervention Description: This is an interrupted time series study where investigators will compare

SUMMARY:
Enhanced interventions are needed to mitigate the impact psychological trauma has on HIV appointment adherence among Black youth with HIV in the Southern United States (U.S.). We will adapt and test an HIV trauma treatment to improve outcomes for both youth with HIV and their HIV care providers in the priority region of Memphis, TN, which houses the third highest rate of new HIV infections, with a third among youth.

DETAILED DESCRIPTION:
Investigators will reduce health disparities among underserved youth in a region with the third highest HIV incidence nationally. Shelby County, Tennessee (TN; Memphis) is a Phase I priority jurisdiction for the U.S. Ending the HIV Epidemic (EHE) initiative, where youth with HIV (YWH) suffer comparatively worse HIV outcomes: half of all YWH in Memphis are appointment non-adherent, representing a major threat to HIV viral suppression, morbidity, and disease transmission. Psychological trauma is a critical and understudied mechanism driving a multitude of HIV-related disparities that will only be eliminated through multi-level solutions. At the patient-level, YWH endure high rates of post-traumatic stress disorder (47%), with adversity due to skin color intensifying experiences among youth; at the personnel-level, repeated trauma exposures associated with HIV care provision contribute to vicarious trauma and degrades professional quality of life. At the clinic-level, trauma sequalae thwart patient-provider relationships and trust, which contributes to treatment fatigue, disengagement, and viral failure. Trauma-Informed care (TIC) is an evidence-based approach that improves multi-level outcomes (e.g., personnel practices, clinic climate, and patient appointment adherence) by ensuring personnel are adequately trained to Recognize and Respond to trauma and Resist Re-traumatization. Though the Memphis EHE plan cites TIC implementation as critical to advancing local goals, the HIV clinic at St. Jude Children's Research Hospital (SJCRH), primary care provider for YWH in the area, has not implemented TIC. Investigators have developed this proposal with SJCRH to support enhanced TIC for youth with HIV (TIC-YH) implementation in their HIV care clinic system. Investigators will conduct a Sequential Transformative Mixed Methods design study through the following three aims: 1) Adapt TIC protocols by incorporating novel contextual components; 2) Implement and assess impact of novel TIC-YH intervention on personnel attitudes, practices, and system culture; and 3) Implement and assess impact of novel TIC-YH on patient HIV appointment adherence and trauma response. This innovative and highly significant research is wholly consistent with NIH high priority areas of research to reduce health disparities in treatment outcomes of those living with HIV and training of workforce conducting high priority HIV-related research. By the end of the 5-year grant period, K01 candidate will have received extensive career development in the areas of implementation science and mixed methods design, enabling the development of a programmatic line of research to advance EHE goals. There is strong rationale to support the current TIC-YH intervention and proposed research methods as meaningful approaches to addressing disparities across a wide range of areas, including chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

* Have a documented HIV+ status and be receiving care from St. Jude HIV clinic
* Be able to participate in English and consent to intervention
* Screen positive for at least one trauma exposure
* Be between the ages of 18-24

Personnel must:

* Be an employee of St. Jude Childrens Research Hospital
* Be at least 18 years of age
* Be able to communicate in English

Exclusion Criteria:

Patients:

• No patients below the age of 18 who cannot communicate in English

Personnel:

* No past employees
* Must be a current St. Jude employee who interfaces with the HIV clinic patients in some capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in knowledge and attitudes of trauma-informed care | This will occur from years 2-3 of the grant (years 1-2 for this clinical trial timeline, as year one is only adaptation and not part of the trial)
  Personnel increases in knowledge and attitudes will be measured via the Trauma-informed Climate Scale (TICS); the Trauma-informed Belief Scale (TIBS); and novel items to accompany the Organizational Trauma Resilience (OTR) Assessment tools listed below.
  TICS is a 5-point Likert scale (1 'Strongly Disagree' to 5 'Strongly Agree), with higher scores indicating higher levels of trauma-informed climate, and ranging from 10-50, with 50 indicating better outcomes.
  TIBS is a 19-item scale measuring trauma-informed beliefs. Higher scores indicate greater outcomes, using a five-point Likert scale (1= Strongly Disagree to 5= Strongly Agree) and scores ranging from 19-95.
  The novel items measure OTR knowledge and attitudes and will be tested for correlation with the TICS and TIBS. There are 29 items: 28 are on a five-point Likert scale and one is on an 8-point slider scale. Scores range from 29-148, with higher scores indicating better outcomes.
Changes in perceived culture of organizational trauma resilience (OTR) in patients | This will occur between years 2-5 of the grant (years 1-4 of the trial)
  Patients will respond to surveys to assess levels of Organizational Trauma Resilience (OTR) in the clinic, using the Organizational Trauma Resilience - Patient Reported Experience Measure, which is a 40-item instrument that has been validated in previous studies and uses a five-point Likert scale. Scores range from 40-200, with higher scores indicating better outcomes.
Changes in perceived culture of organizational trauma resilience (OTR) in personnel | This will occur between years 2-5 of the grant (years 1-4 of the trial)
  Personnel will respond to surveys to assess levels of Organizational Trauma Resilience (OTR) in the clinic, using the Organizational Trauma Resilience Assessment. This is a 40-item instrument that has been validated in previous studies and uses a five-point Likert scale. Scores range from 40-200, with higher scores indicating better outcomes.
Number of patients adherent to medical appointment | This will occur in years 3-5 of the study (years 2-4 of the trial)
  Patient appointment adherence will be tracked (missed/attended versus scheduled appointments)
Changes in trauma response: PTSD | This will occur in years 3-5 of the study (years 2-4 of the trial)
  Patients will be assessed for post-traumatic stress symptoms over time using the Short Post-Traumatic Stress Disorder Rating Interview scale (SPRINT). This is an 8-item instrument measuring PTSD symptoms on a five-point Likert scale (0= Not at all and 4= Very Much), with higher scores indicating worse outcomes. The possible range of scores is 0-32.
Changes in trauma response: Complex PTSD | This will occur in years 3-5 of the study (years 2-4 of the trial)
  Patients will be assessed for post-traumatic stress symptoms over time using the International Trauma Questionnaire. This is an 18-item scale, using a five-point Likert scoring (0=Not at all, 5= Extremely), with a possible range of scores as 0-72 and higher scores as worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Jude Childrens Research Hospital, Memphis, Tennessee, United States

DOCUMENTS (3):
  • Study Protocol (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT07137026/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT07137026/SAP_001.pdf
  • Informed Consent Form (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT07137026/ICF_002.pdf